CLINICAL TRIAL: NCT06162351
Title: A Phase II Study to Evaluate the Efficacy and Toxicities of PLX038, in Patients With Locally Advanced or Metastatic Triple-negative Breast Cancer
Brief Title: A Study to Evaluate the Efficacy and Toxicities of PLX038, in Patients With Locally Advanced or Metastatic Triple-negative Breast Cancer
Acronym: TOPOLOGY
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No signal of significant toxicity and no signal of activity in the population of the TOPOLGY study
Sponsor: Institut Curie (Other)
Collaborators: ProLynx LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC 2020-16
Record Dates: First submitted 2023-11-13; First posted 2023-12-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Breast; Cancer
Keywords: Pretreated; Metastatic; Locally; Advanced triple negative
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Single arm phase II study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm: treatment with PLX038 (Experimental): Patients will be treated at a dose of 1730mg/m2 IV infusion on Day 1 of each cycle Q3W (every 21 days, 1 cycle = 1 injection).
  Interventions: Drug: PLX038

INTERVENTIONS:
Drug: PLX038 — Study treatment will be at a dose of 1730mg/m2 IV infusion on Day 1 of each cycle Q3W (every 21 days, 1 cycle = 1 injection).
  Patients with a clinical benefit could be treated as long as study is ongoing. Patients are followed from inclusion until documented disease progression, withdrawal of consent, or death.

SUMMARY:
Single arm phase II study for with primary objective to evaluate the efficacy of PLX038 on response rate for patients with pretreated, metastatic or locally advanced triple negative breast cancer.

DETAILED DESCRIPTION:
This is an open label, multi-centric phase II study designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and efficacy of PLX038 in locally-advanced or metastatic TNBC. Patient must have received prior therapy (administered in the neoadjuvant, adjuvant and/or metastatic setting) with chemotherapy by an anthracycline, taxane and sacituzumab-govitecan (unless not medically appropriate or contraindicated for the patient) and received a minimum of two prior cytotoxic chemotherapy regimens for locally advanced or metastatic breast cancer.

Patients will be treated at a dose of 1730mg/m2 IV infusion on Day 1 of each cycle Q3W (every 21 days, 1 cycle = 1 injection).

All included patients will receive PLX038 as single agent as long as study is ongoing or until progression of disease, unacceptable toxicity, patient withdrawal of consent, Investigator decision, lost to follow-up, death, patient non-compliance, or study termination by Sponsor.

Tumor assessments must be performed according to the RECIST V1.1 criteria at inclusion and every 8 weeks (± 7 days) from inclusion until documented disease progression, withdrawal of consent, or death. Radiographic measurements must be performed to the RECIST specifications.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with the protocol and provide written informed consent prior to study-specific screening procedures.
* Age ≥ 18 years.
* Females and males with cytologically or histologically confirmed breast carcinoma (either the primary or metastatic lesions).
* Locally advanced or metastatic disease that is not amenable to curative treatment.
* Triple negative breast cancer (both ER and PR <10%, HER2-negative or HER2-low).
* Measurable disease (per RECIST version 1.1).
* Prior therapy (administered in the neoadjuvant, adjuvant and/or metastatic setting) with chemotherapy by an anthracycline, taxane and sacituzumab-govitecan (unless not medically appropriate or contraindicated for the patient).
* Received a minimum of two prior cytotoxic chemotherapy regimens for locally advanced or metastatic breast cancer.
* Patients with known gBRCA mutations must have received a PARP inhibitor in the metastatic setting.
* Patients whose cancer has a CPS score ≥10 must have received prior pembrolizumab unless (i) contra-indicated (ii) CPS score or pembrolizumab not available at time of first line treatment start.
* Resolution of chemotherapy and radiation therapy related toxicities to NCI-CTCAE version 5.0 Grade 1 or lower severity, except for stable sensory neuropathy (≤ Grade 2), alopecia (any grade), presence of clinically managed chronic autoimmune AEs from prior immune therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function (obtained within 14 days prior to treatment start) as evidenced by:

  i. Absolute neutrophil count (ANC) ≥ 1.5 X 109/L; ii. Hemoglobin (Hgb) ≥ 9 g/dL; iii. Platelet count ≥ 100 X 109/L; iv. Bilirubin ≤ 1.5 X upper limit of normal (ULN), except for patients with a documented history of Gilbert's disease (≤ 2 X ULN); v. Alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ 2.5 X ULN (for patients with liver metastases ≤ 5 X ULN); vi. Alkaline phosphatase (AP) ≤ 3 X ULN (for patients with liver metastases, ≤ 5 X ULN); vii. Serum creatinine ≤ 1.5 mg/dL (133 μmol/L) or calculated creatinine clearance ≥ 50 mL/min (using Cockcroft-Gault formula); viii. Women of childbearing potential (WCBP): negative serum pregnancy test.
* Patients covered by social security or health insurance in compliance with the national legislation relating to biomedical research.

Exclusion Criteria:

* Patients who had a last dose of IV chemotherapy within 21 days, last dose of oral cytotoxic chemotherapy, radiotherapy, biological therapy, or investigational therapy within 14 days prior to treatment start.
* Patients who had any major surgery within 28 days prior to inclusion.
* Patients with chronic inflammatory bowel disease and/or bowel obstruction.
* Concomitant use of other agents for the treatment of cancer or any investigational agent(s).
* Brain metastases, unless local therapy was completed and use of corticosteroids for this indication discontinued for at least 3 weeks prior to inclusion. Signs or symptoms of brain metastases must be stable for at least 28 days prior to inclusion. No known progression of brain metastases (by imaging as assessed by RECIST) can have occurred. Patients with leptomeningeal disease or meningeal carcinomatosis are excluded.
* Women who are either pregnant, lactating, planning to get pregnant.
* Patients receiving pharmacotherapy for hepatitis B or C, tuberculosis, or HIV.
* Patients with known liver disease diagnosed with Child-Pugh A or higher cirrhosis.
* Prior stage III or IV malignancy (other than breast cancer).
* Severe/uncontrolled intercurrent illness within the previous 28 days prior to inclusion.
* Significant known cardiovascular impairment (NYHA CHF > grade 2, unstable angina, myocardial infarction within the previous 6 months prior to inclusion, or existing unstable cardiac arrhythmia).
* Any other significant medical, psychological, social or geographic conditions that in the opinion of the Investigator would impair study participation or cooperation.
* Patients deprived of their liberty or under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Best tumor response | 24 weeks
  Best tumor response (defined as PR or CR in the first 6 months of treatment, assessed by investigators per RECIST v1.1 criteria).

SECONDARY OUTCOMES:
Time to response (TTR) | Until 24 months
  Time to response is defined as the time from inclusion to the first objective tumor response and will be estimated using Kaplan-Meier method
SAEs (all grade, per NCI-CTCAE v5.0) | Until 30 days after the last dose of IMP (24 months + 30 days)
  Serious adverse events (SAEs)according to NCI CTCAE v5.0, by grade and their relationship to PLX038
Correlation between PLX038 efficacy and homologous recombination (HR) defect (assessed by HR genes mutational status and BCRAness phenotype) | Until 24 months
  Incidence of efficacy of PLX038 in pre-defined biomarker subgroups (BRCAness)
PK analysis | Until 24 months
  Maximum Plasma Concentration effect of PLX038
Duration of Response (DoR) | Until 24 months
  DoR is defined as the time from the first documented PR or CR until the date of disease progression or the date of death. DoR will be computed using Kaplan-Meier
Progression free survival (PFS) | Until 24 months
  PFS is defined as the time from inclusion to progression (per RECIST 1.1) or death, among included patients
Overall Survival (OS) | Until 24 months
  PFS is defined as the time from inclusion to the first event among progression and death. OS is defined in the same way but only death is taken into account.
AEs | Until 30 days after the last dose of IMP (24 months + 30 days)
  Adverse events (AEs) according to NCI CTCAE v5.0, by grade and their relationship to PLX038
Correlation between PLX038 efficacy and homologous recombination (HR) defect, replication stress-related biomarkers such as SFLN11 expression | Until 24 months
  Incidence of efficacy of PLX038 in pre-defined biomarker subgroups (SLFN11 expression)
Correlation between PLX038 efficacy and homologous recombination (HR) defect replication stress-related biomarkers such as RB1 loss | Until 24 months
  Incidence of efficacy of PLX038 in pre-defined biomarker subgroups (RB1 loss)
PD analysis | Until 24 months
  Maximum Plasma Concentration of effect of PLX038

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut Curie, Paris
  - Institut Curie, Saint-Cloud

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).